CLINICAL TRIAL: NCT07185204
Title: Postpartum Preeclampsia Early Detection and Treatment: Using Biomarkers to Implement Risk-stratified Intervention (Nepal Pilot Randomized Controlled Trial)
Brief Title: Postpartum Preeclampsia Early Detection and Treatment: Nepal Pilot Study
Acronym: PREDiCT-NPL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Dhulikhel Hospital (Other)
Responsible Party: Principal Investigator, Anna Palatnik, MD, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO00056073
Record Dates: First submitted 2025-06-30; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Postpartum Preeclampsia
Keywords: Preeclampsia; Hypertension; Pregnancy; Postpartum
MeSH Terms: conditions — Pre-Eclampsia; Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-risk Intervention (Experimental): Participants with high-risk sFlt-1/PlGF ratio randomized to early detection and management of postpartum preeclampsia with remote blood pressure monitoring, education, and dispensing antihypertensive medication (nifedipine ER) for outpatient management of asymptomatic, mild range BP.
  Interventions: Other: Early detection and management of postpartum preeclampsia bundle
- High-Risk Control (No Intervention): Participants with high-risk sFlt-1/PlGF ratio randomized to standard postpartum care.
- Low-risk Control (No Intervention): Participants with low-risk sFlt-1/PlGF ratio will not be randomized, but will remain enrolled to assess the exploratory outcome of biomarker predictive ability.

INTERVENTIONS:
Other: Early detection and management of postpartum preeclampsia bundle — Remote blood pressure monitoring, education, and dispensing antihypertensive medication (nifedipine ER) for outpatient management of asymptomatic, mild range BP.
  Arms: High-risk Intervention

SUMMARY:
The goal of this study is to address the significant morbidity associated with preeclampsia diagnosed after delivery. All participants will undergo biomarker evaluation with soluble fms-like tyrosine kinase-1 and placental growth factor (sFlt-1/PlGF) ratio testing before delivery to assess the predictive ability of these biomarkers with new-onset postpartum preeclampsia. High-risk participants will be randomized to a bundle of care strategies aimed at early detection and management of postpartum preeclampsia.

DETAILED DESCRIPTION:
This is a pilot randomized controlled trial of 60 normotensive, pregnant patients randomized to early monitoring and management for postpartum preeclampsia after biomarker evaluation with sFlt-1/PlGF ratio. After obtaining informed consent, participants will undergo preeclampsia risk assessment using sFlt-1/PlGF ratio testing prior to delivery. Patients with a low risk ratio will receive routine postpartum care. Patients with a high risk ratio will be randomized 1:1 to the intervention bundle focused on early detection and management of postpartum preeclampsia versus routine postpartum care. The intervention bundle will include remote blood pressure monitoring, education, and dispensing antihypertensive medication (nifedipine ER) for outpatient management of asymptomatic, mild-range BP. The primary outcome is the feasibility of all study procedures, measured by recruitment, retention, adherence, and acceptability. The secondary outcome is to assess the effect of early monitoring and management of postpartum preeclampsia on the composite outcome of hypertension requiring in-person medical evaluation and hypertension-related morbidity. Finally, the exploratory outcome is the predictive ability of sFlt-1/PlGF ratio of de novo postpartum preeclampsia in antenatally normotensive patients who are at risk for HDP based on ACOG/USPSTF criteria. Data on primary and secondary outcomes will be collected from both randomized groups and the non-randomized group with low-risk sFlt-1/PlGF ratio to determine the predictive capability of the test in the postpartum period.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients ≥ 36 weeks gestation without major fetal anomalies
* Age ≥ 18 years
* Admitted for labor at Dhulikhel Hospital, or intend to deliver at Dhulikhel Hospital
* At risk for preeclampsia, using the Clinical Risk Assessment for Preeclampsia according to ACOG and USPSTF

  * 1 or more high risk factors:

    * History of preeclampsia
    * Type 1 or 2 diabetes
    * Multifetal gestation?
    * Renal disease
    * Autoimmune disease
  * 2 or more moderate risk factors:

    * Nulliparity
    * BMI > 30
    * First-degree relative with a history of preeclampsia
    * African American race
    * Low socioeconomic status
    * Age > 35 years
    * History of low birthweight or small for gestational age
    * Previous adverse pregnancy outcome
    * Interpregnancy interval > 10 years

Exclusion Criteria:

* Antenatal hypertensive disorder of pregnancy diagnosis, including gestational hypertension, preeclampsia, eclampsia, or HELLP syndrome, according to ACOG guidelines
* Chronic hypertension, according to ACOG guidelines
* Known allergy or contraindication to nifedipine
* Inability or unwillingness to provide informed consent
* Two or more blood pressures with an SBP ≥140 or DBP ≥90 after consent and prior to sFlt-1/PlGF testing (screen failure criteria)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Study feasibility | 1 year
  Assess study feasibility as measured by retention rate.

SECONDARY OUTCOMES:
Composite outcome of hypertension-related healthcare utilization and morbidity. | 4 weeks postpartum
  Assess the effect of early monitoring and management of postpartum preeclampsia on the incidence of a composite outcome including hypertension requiring in-person medical evaluation and hypertension-related morbidity.
Predictive ability of sFlt-1/PlGF ratio for de novo postpartum preeclampsia | 2 weeks postpartum
  Assess the sFlt-1/PlGF ratio predictive ability of de novo postpartum preeclampsia in antenatally normotensive patients.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Palatnik, MD, Principal Investigator — Medical College of Wisconsin
Locations (2):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States
- Dhulikhel Hospital, Dhulikhel, Nepal

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared since this is a pilot study with very small sample sizes in each randomization group.